CLINICAL TRIAL: NCT06399263
Title: Study of Psilocybin for Anorexia in Young Adults
Acronym: SPANYA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marissa Raymond-Flesch, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Marissa Raymond-Flesch, MD, MPH, Professor, Pediatrics, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-39236
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin Therapy (Experimental): The psilocybin therapy will include three preparatory sessions, psilocybin dosing session one (20mg), two integration sessions, psilocybin dosing session two (up to 25mg), and four final integration sessions
  Interventions: Drug: Psilocybin; Behavioral: Preparation and Integration Sessions

INTERVENTIONS:
Drug: Psilocybin — The psilocybin will include two dose administration sessions, first a 20mg administration, and second an administration of up to 25mg.
  Other Names: PEX010
Behavioral: Preparation and Integration Sessions — The psilocybin therapy will include three preparatory sessions, two dose A integration sessions, and four final integration sessions.
  Other Names: Psilocybin Therapy

SUMMARY:
This is a single site trial of psilocybin therapy for the treatment of refractory Anorexia Nervosa in young adults. The psilocybin therapy will include three preparatory sessions, psilocybin dosing session one (20mg), two integration sessions, psilocybin dosing session two (up to 25mg), and four final integration sessions. Eating disorder symptoms will be measured pre and post treatment. One to two family member(s) of each young adult participant will be enrolled in the study. One of which will be required to attend a portion of two preparatory sessions and a portion of two integration sessions and receive psychoeducation about supporting the young adult participant through preparation and integration for psilocybin therapy. Investigators hypothesize that psilocybin will increase cognitive flexibility and that this increase will predict long-term changes in cognitive rigidity, habitual eating, and exercise behaviors in patients with Anorexia Nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent.
* Between 18 and 25 years old at time of screening.
* Meets Diagnostic and Statistical Manual (DSM-5) criteria for any type of Anorexia Nervosa
* Currently experiencing symptoms of Anorexia Nervosa
* Comfortable reading and writing in English
* Have no anticipated changes in medication or surgical procedures for trial duration
* Commit to attend all in-person and remote study visits and participate in all data collection procedures
* Able to identify one or two family members or close friends to co-enroll in the study, who will be required to participate in select therapy sessions.
* Agree to use a highly effective form of contraception for two weeks prior to starting the study and one month after finishing the study.
* Agree that for one week preceding each psilocybin session, they will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the research team. Exceptions will be evaluated by the research team and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Agree to consume approximately the same amount of caffeine-containing beverages (e.g., coffee, tea) that they usually consume before arriving at the research unit on the mornings of psilocybin administration sessions. If the young adult participant does not routinely consume caffeinated beverages, they must agree not to do so prior to psilocybin administration sessions.

Exclusion Criteria:

* Current known pregnancy or positive pregnancy test at any time during the study
* Personal history of bipolar disorder, or psychotic disorder verified by the Structured Clinical Interview for DSM-5 (SCID) and medical history at screening
* Body Mass Index less than 12 at screening
* Unstable vital signs including Blood Pressure, Heart Rate, or Temperature
* Abnormal Safety Labs including sodium, potassium, magnesium, phosphorus, creatinine, estimated Glomerular Filtration Rate, Aspartate Transferase, Alanine Transaminase
* Electrocardiogram abnormalities
* Hospitalization or participation in a residential program for more than 2 of the past 4 weeks at the time of screening.
* Unwilling to abstain from alcohol, Cannabidiol (CBD), tetrahydrocannabinol (THC), marijuana, and illicit drug use for 48 hours pre and post psilocybin dosing days and abstain from nicotine for 10 hours pre and post psilocybin dosing.
* Positive urine toxicology testing for amphetamines, benzodiazepines, cocaine, cannabis, 3,4-Methylenedioxymethamphetamine (MDMA), and opioids (including methadone and buprenorphine) on the morning of either psilocybin administration session.
* History of cardiovascular disease
* Uncontrolled endocrine conditions, including diabetes, hyper or hypothyroidism
* Significant and uncontrolled gastrointestinal illness at the discretion of the investigator
* Significant and uncontrolled neurological disease including uncontrolled seizure disorder at the discretion of the investigator
* Use of any prohibited concomitant medications or inability or unwillingness to discontinue according to the study's prescribed medication taper or tapering with the participants primary prescriber.
* Needle phobia.
* Simultaneous enrollment in another clinical trial.
* Pregnant or Breast feeding.
* Allergy or intolerance to any of the materials contained in the drug product
* History of severe reaction to psychedelics at the discretion of the investigators.
* High risk of self-harm/suicide
* Mental health condition that will prevent engagement with the treatment team.
* Unwilling or unable to participate in the treatment protocol as planned, including hydration with sports drinks on dosing days.
* If any study physician feels that it would be unsafe to continue for any mental, physical or other reason

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination (EDE) | Baseline, 28 days, 90 days, 365 days
  The EDE assess eating disorder behaviors and attitudes though an interviewer administered questionnaire. It provides 4 subscale scores (Restraint, Eating Concern, Shape Concern and Weight Concern). Score range from 0 to 6 and are averaged to calculate a global score. Higher scores indicate increased eating disorder thoughts and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Raymond-Flesch, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://redcap.ucsf.edu/surveys/?s=AK99FE8XM4YRTYMY